CLINICAL TRIAL: NCT01774487
Title: A Phase II Trial of Pentoxifylline in Newly-Diagnosed Biliary Atresia
Brief Title: Pentoxifylline Therapy in Biliary Atresia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Target enrollment was not reached because the medication, pentoxifylline, has a taste that is not well tolerated by infants. The study team decided to end the study before meeting the enrollment goal because of the medication taste.
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Sanjiv Harpavat, Assistant Professor, Department of Pediatrics, Division of Gastroenterology, Hepatology, and Nutrition, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-31387
Record Dates: First submitted 2013-01-22; First posted 2013-01-24 (Estimated); Results first posted 2023-10-12 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Biliary Atresia
Keywords: Biliary Atresia; Pentoxifylline; Trental; Serum bilirubin; Conjugated bilirubin; Liver transplantation; Fibrosis
MeSH Terms: conditions — Biliary Atresia; Fibrosis | interventions — Pentoxifylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pentoxifylline (Experimental): All newly-diagnosed biliary atresia patients fulfilling the study's inclusion criteria will receive oral pentoxifylline, 20 mg/kg/day divided in three doses for a total of 90 days.
  The hospital pharmacy will create a 20 mg/ml oral pentoxifylline solution using 400 mg pentoxifylline tablets and established compounding recipes.
  Interventions: Drug: Pentoxifylline

INTERVENTIONS:
Drug: Pentoxifylline — 20 mg/kg/day divided in 3 doses, given orally for 90 days
  Other Names: Trental

SUMMARY:
The purpose of this study is to determine whether pentoxifylline reduces liver damage in infants with biliary atresia.

DETAILED DESCRIPTION:
Biliary atresia (BA) is a devastating liver disease of infancy of unknown etiology, characterized by bile duct obstruction, live fibrosis, and cirrhosis. BA has no known medical treatments. The only proven treatment is a surgical portoenterostomy (the Kasai procedure, or KP) which can achieve bile drainage and improve outcomes in some cases. The KPs success is variable depending on several factors including age of the infant, experience of the surgeon, and extent of liver fibrosis at the time of KP.

In this study, the investigators conduct a phase II trial of a potential new medical therapy for BA: pentoxifylline (PTX). PTX is a methylxanthine derivative closely related to caffeine that has been used safely in infants with other diseases such as sepsis. In adults, PTX has been shown to have a number of properties beneficial to the liver, including preventing liver fibrosis, improving liver regeneration, and reducing cirrhosis-related complications.

The trial's objective is to determine whether PTX has sufficient biological activity against BA to warrant further study. PTX will be administered orally for 90 days as an adjunct to standard therapy (i.e. KP if appropriate). The primary outcome will measure the change in serum conjugated bilirubin levels after 90 days. Secondary outcomes include changes in body weight, serum markers, liver imaging, and time to liver transplant in infants with BA.

ELIGIBILITY:
Inclusion Criteria:

* 0-180 days old
* Diagnosed with biliary atresia through liver biopsy and/or intra-operative cholangiogram
* No previous Kasai portoenterostomy performed at another institution
* Able to take medications orally
* Legal guardian signs consent after understanding risks and investigational nature of study

Exclusion Criteria:

* Infants greater than 180 days old
* Infants receiving a Kasai portoenterostomy at another institution
* Infants unable to take medications orally

Max Age: 180 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2013-02-04 (Actual); Primary Completion 2018-02-07 (Actual); Study Completion 2023-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjiv Harpavat, MD PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital and Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
The data for subjects will be shared in aggregate.

REFERENCES:
- [Background] Perlmutter DH, Shepherd RW. Extrahepatic biliary atresia: a disease or a phenotype? Hepatology. 2002 Jun;35(6):1297-304. doi: 10.1053/jhep.2002.34170. No abstract available. PMID 12029613
- [Background] Sokol RJ, Shepherd RW, Superina R, Bezerra JA, Robuck P, Hoofnagle JH. Screening and outcomes in biliary atresia: summary of a National Institutes of Health workshop. Hepatology. 2007 Aug;46(2):566-81. doi: 10.1002/hep.21790. PMID 17661405
- [Background] Garcia AV, Cowles RA, Kato T, Hardy MA. Morio Kasai: a remarkable impact beyond the Kasai procedure. J Pediatr Surg. 2012 May;47(5):1023-7. doi: 10.1016/j.jpedsurg.2012.01.065. PMID 22595595
- [Background] Shneider BL, Brown MB, Haber B, Whitington PF, Schwarz K, Squires R, Bezerra J, Shepherd R, Rosenthal P, Hoofnagle JH, Sokol RJ; Biliary Atresia Research Consortium. A multicenter study of the outcome of biliary atresia in the United States, 1997 to 2000. J Pediatr. 2006 Apr;148(4):467-474. doi: 10.1016/j.jpeds.2005.12.054. PMID 16647406
- [Background] Weerasooriya VS, White FV, Shepherd RW. Hepatic fibrosis and survival in biliary atresia. J Pediatr. 2004 Jan;144(1):123-5. doi: 10.1016/j.jpeds.2003.09.042. PMID 14722530
- [Background] Zhang D, Jiang H, Wang Y, Ma J. Pentoxifylline inhibits hepatic stellate cells proliferation via the Raf/ERK pathway. APMIS. 2012 Jul;120(7):572-81. doi: 10.1111/j.1600-0463.2011.02868.x. Epub 2012 Jan 19. PMID 22716212
- [Background] Andrade Wde C, Tannuri U, da Silva LF, Alves VA. Effects of the administration of pentoxifylline and prednisolone on the evolution of portal fibrogenesis secondary to biliary obstruction-an experimental study in growing animals. J Pediatr Surg. 2009 Nov;44(11):2071-7. doi: 10.1016/j.jpedsurg.2009.05.020. PMID 19944210
- [Background] Zein CO, Yerian LM, Gogate P, Lopez R, Kirwan JP, Feldstein AE, McCullough AJ. Pentoxifylline improves nonalcoholic steatohepatitis: a randomized placebo-controlled trial. Hepatology. 2011 Nov;54(5):1610-9. doi: 10.1002/hep.24544. Epub 2011 Aug 24. PMID 21748765
- [Background] Petrowsky H, Breitenstein S, Slankamenac K, Vetter D, Lehmann K, Heinrich S, DeOliveira ML, Jochum W, Weishaupt D, Frauenfelder T, Graf R, Clavien PA. Effects of pentoxifylline on liver regeneration: a double-blinded, randomized, controlled trial in 101 patients undergoing major liver resection. Ann Surg. 2010 Nov;252(5):813-22. doi: 10.1097/SLA.0b013e3181fcbc5e. PMID 21037437
- [Background] Lebrec D, Thabut D, Oberti F, Perarnau JM, Condat B, Barraud H, Saliba F, Carbonell N, Renard P, Ramond MJ, Moreau R, Poynard T; Pentocir Group. Pentoxifylline does not decrease short-term mortality but does reduce complications in patients with advanced cirrhosis. Gastroenterology. 2010 May;138(5):1755-62. doi: 10.1053/j.gastro.2010.01.040. Epub 2010 Jan 25. PMID 20102716
- [Background] Haque KN, Pammi M. Pentoxifylline for treatment of sepsis and necrotizing enterocolitis in neonates. Cochrane Database Syst Rev. 2011 Oct 5;(10):CD004205. doi: 10.1002/14651858.CD004205.pub2. PMID 21975745
- [Background] Superina R, Magee JC, Brandt ML, Healey PJ, Tiao G, Ryckman F, Karrer FM, Iyer K, Fecteau A, West K, Burns RC, Flake A, Lee H, Lowell JA, Dillon P, Colombani P, Ricketts R, Li Y, Moore J, Wang KS; Childhood Liver Disease Research and Education Network. The anatomic pattern of biliary atresia identified at time of Kasai hepatoportoenterostomy and early postoperative clearance of jaundice are significant predictors of transplant-free survival. Ann Surg. 2011 Oct;254(4):577-85. doi: 10.1097/SLA.0b013e3182300950. PMID 21869674
- [Background] Simon R. Optimal two-stage designs for phase II clinical trials. Control Clin Trials. 1989 Mar;10(1):1-10. doi: 10.1016/0197-2456(89)90015-9. PMID 2702835
- [Background] Best BM, Burns JC, DeVincenzo J, Phelps SJ, Blumer JL, Wilson JT, Capparelli EV, Connor JD; Pediatric Pharmacology Research Unit Network. Pharmacokinetic and tolerability assessment of a pediatric oral formulation of pentoxifylline in kawasaki disease. Curr Ther Res Clin Exp. 2003 Feb;64(2):96-115. doi: 10.1016/S0011-393X(03)00018-3. PMID 24944359
- [Background] Davenport M, Caponcelli E, Livesey E, Hadzic N, Howard E. Surgical outcome in biliary atresia: etiology affects the influence of age at surgery. Ann Surg. 2008 Apr;247(4):694-8. doi: 10.1097/SLA.0b013e3181638627. PMID 18362634

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All newly-diagnosed biliary atresia patients fulfilling the study's inclusion criteria (those who received the Kasai portoenterostomy are in Group 1 and those diagnosed too late for the Kasai portoenterostomy are in Group 2)
Groups:
- Pentoxifylline - Group 1 (Treatment Starts 3-5 Days After Kasai Portoenterostomy); Pentoxifylline - Group 2 (Patient Diagnosed Too Late for Kasai Portoenterostomy): All newly-diagnosed biliary atresia patients fulfilling the study's inclusion criteria will receive oral pentoxifylline, 20 mg/kg/day divided in three doses for a total of 90 days.
  The hospital pharmacy will create a 20 mg/ml oral pentoxifylline solution using 400 mg pentoxifylline tablets and established compounding recipes.
  Pentoxifylline: 20 mg/kg/day divided in 3 doses, given orally for 90 days
Period: Overall Study
Arm/Group | Pentoxifylline - Group 1 (Treatment Starts 3-5 Days After Kasai Portoenterostomy) | Pentoxifylline - Group 2 (Patient Diagnosed Too Late for Kasai Portoenterostomy)
Started | 12 | 5
Completed | 8 | 1
Not Completed | 4 | 4
Not completed — Did not tolerate taste | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Pentoxifylline Group 1; Pentoxifylline Group 2: All newly-diagnosed biliary atresia patients fulfilling the study's inclusion criteria will receive oral pentoxifylline, 20 mg/kg/day divided in three doses for a total of 90 days.
  The hospital pharmacy will create a 20 mg/ml oral pentoxifylline solution using 400 mg pentoxifylline tablets and established compounding recipes.
  Pentoxifylline: 20 mg/kg/day divided in 3 doses, given orally for 90 days
- Total: Total of all reporting groups
Arm/Group | Pentoxifylline Group 1 | Pentoxifylline Group 2 | Total
Number analyzed (Participants) | 12 | 5 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 5 | 17
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: days] — Age at Kasai portoenterostomy (Group 1) or Age at Presentation (Group 2)
  days | 49 (26) | 120 (30) | 69 (42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 2 | 10
  Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 7
  Not Hispanic or Latino | 7 | 3 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 9 | 4 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Normal Serum Conjugated Bilirubin Levels 12 Weeks After Starting PTX (Pentoxifylline) Therapy
Description: The investigators will track the serum conjugated bilirubin (CB) levels over the course of therapy in patients receiving 90 days of PTX (this laboratory test is drawn as part of routine care). Normal CB is 0.0-0.3 mg/dL, with a higher number of patients meeting this indicating a better outcome.
Time Frame: 12 weeks after starting therapy
Measure: Count of Participants; unit: Participants
Groups:
- Pentoxifylline - Group 1: Infants receiving the Kasai portoenterostomy (KP) will be given PTX for 12 weeks, and the number whose CB levels return to normal (0.0-0.3 mg/dL) will be calculated. Historically, ~60% of such infants have normal CB levels after 12 weeks. The study will determine whether PTX improves this percentage.
- Pentoxifylline - Group 2: For Group 2: Infants not receiving the KP will be given PTX for 12 weeks, and the number whose CB levels stabilize (within 10% of starting level) will be calculated. Historically, ~10% of such infants have stable CB levels after 12 weeks. The study will determine whether PTX improves this percentage.
Arm/Group | Pentoxifylline - Group 1 | Pentoxifylline - Group 2
Number analyzed (Participants) | 8 | 1
Participants | 6 | 0

2. Secondary Outcome: Number of Participants Achieving Zero or Positive Weight Z-scores 12 Weeks After Starting PTX Therapy
Description: The investigators will track the weight of patients over the course of therapy in patients receiving 90 days of PTX (this is recorded as part of routine clinical care). The weight will then be compared to standards to calculate a z-score. Normal weight Z-score is greater than or equal to 0, with a higher number of patients meeting this indicating a better outcome.
Time Frame: 12 weeks after starting therapy
Measure: Count of Participants; unit: Participants
Groups:
- Pentoxifylline - Group 1: Infants receiving the KP will be given PTX for 12 weeks, and the number with weight z-scores greater than or equal to 0 on the World Health Organization (WHO) growth chart will be counted.
- Group 2: For Group 2: Infants not receiving the KP will be given PTX for 12 weeks, and the number with weight z-scores greater than or equal to 0 on the WHO growth chart will be counted.
Arm/Group | Pentoxifylline - Group 1 | Group 2
Number analyzed (Participants) | 8 | 1
Participants | 0 | 0

3. Secondary Outcome: Alanine Amino Transferase (ALT) Levels at 2 Years of Life
Description: The investigators will record the ALT levels at age two years, in patients who had previously been treated with PTX therapy and still have their native liver. Range of normal values: 14-45 U/L, with a higher level indicating a worse outcome.
Time Frame: 2 years of age
Population: No patient in Group 2 survived with their native liver to 2 years of age.
Measure: Mean (Standard Deviation); unit: U/L
Groups:
- Pentoxifylline - Group 1: Infants receiving the KP will be given PTX for 12 weeks, and the ALT levels at 2 years of age will be calculated and reported as average and standard deviation.
- Pentoxifylline - Group 2: Infants not receiving the KP will be given PTX for 12 weeks, and the ALT levels at 2 years of age will be calculated and reported as average and standard deviation.
Arm/Group | Pentoxifylline - Group 1 | Pentoxifylline - Group 2
Number analyzed (Participants) | 6 | 0
U/L | 160 (122) |

4. Secondary Outcome: Spleen Size at 2 Years of Age
Description: The investigators will measure spleen size by ultrasound at 2 years of age, in patients who had received PTX therapy earlier and still have their native liver. "Normal" spleen size range (10th-90th percentile) at this age is 6.4-8.6 cm, with a value exceeding this range indicating a worse outcome.
Time Frame: 2 years of age
Population: No patient in Group 2 survived with their native liver to 2 years of age.
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Pentoxifylline - Group 1: Infants receiving the KP will be given PTX for 12 weeks, and the spleen size will be measured at 2 years.
- Pentoxifylline - Group 2: Infants not receiving the KP will be given PTX for 12 weeks, and the spleen size will be measured at 2 years.
Arm/Group | Pentoxifylline - Group 1 | Pentoxifylline - Group 2
Number analyzed (Participants) | 4 | 0
cm | 10.0 (1.8) |

5. Secondary Outcome: Time to Liver Transplant
Description: The investigators will track time to liver transplant. The shorter time to liver transplant indicates a worse outcome.
Time Frame: Baseline and up to two years after therapy finishes
Measure: Mean (Standard Deviation); unit: days
Groups:
- Pentoxifylline - Group 1: Infants receiving the KP will be given PTX for 12 weeks, and, for those undergoing transplant in the first 2 years of life, the age at transplant will be recorded.
- Pentoxifylline - Group 2: Infants not receiving the KP will be given PTX for 12 weeks, and, for those undergoing transplant in the first 2 years of life, the age at transplant will be recorded.
Arm/Group | Pentoxifylline - Group 1 | Pentoxifylline - Group 2
Number analyzed (Participants) | 2 | 1
days | 317 (95) | 273 (NA) — The is only 1 patient in Group 2

6. Secondary Outcome: Platelet Levels at 2 Years of Life
Description: The investigators will record platelet levels at age two years, in patients who had previously been treated with PTX therapy and still have their native liver. Scale 189-403*10^3 Platelets/μL, with a lower level indicating a worse outcome.
Time Frame: 2 years of age
Population: No patient in Group 2 survived with their native liver to 2 years of age.
Measure: Mean (Standard Deviation); unit: 10^3 Platelets/μL
Groups:
- Pentoxifylline - Group 1: Infants receiving the KP will be given PTX for 12 weeks, and platelet levels at 2 years of age will be calculated and reported as average and standard deviation
- Pentoxifylline - Group 2: Infants not receiving the KP will be given PTX for 12 weeks, and platelet levels at 2 years of age will be calculated and reported as average and standard deviation.
Arm/Group | Pentoxifylline - Group 1 | Pentoxifylline - Group 2
Number analyzed (Participants) | 6 | 0
10^3 Platelets/μL | 208 (102) |

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data was collected for 12 weeks after the Kasai portoenterostomy (duration of time when patient received medication during the study). Note: Some secondary outcomes were collected at age 2 years, but AEs (included all-cause mortality) were collected for 12 weeks after Kasai portoenterostomy to capture those AEs that could possibly be related to treatment.
Description: 1. AEs related to the progression of biliary atresia (BA) include (elevated liver function tests, thrombocytopenia, ascites, cholangitis, failure to thrive, bile leak)
  2. AEs related to PTX, as previously reported, include: vomiting/spitting out medications, abdominal discomfort, cough, anemia with new heart murmur, rhinorrhea, diaper rash, irritability, and temporary hearing loss.
  Serious AEs were any AEs requiring hospitalization.
Arm/Group | Pentoxifylline - Group 1 (Treatment Starts 3-5 Days After Kasai Portoenterostomy) | Pentoxifylline - Group 2 (Patient Diagnosed Too Late for Kasai Portoenterostomy)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/1
Serious Adverse Events (participants affected / at risk) | 6/8 | 1/1
Other Adverse Events (participants affected / at risk) | 4/8 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pentoxifylline - Group 1 (Treatment Starts 3-5 Days After Kasai Portoenterostomy) (N=8) | Pentoxifylline - Group 2 (Patient Diagnosed Too Late for Kasai Portoenterostomy) (N=1)
Failure to thrive (Gastrointestinal disorders) | 3 (5) | 1 (5) — Hospital admission for nutrition optimization (expected with biliary atresia)
Cholangitis (Hepatobiliary disorders) | 2 (3) | 0 (0) — Hospital admission for cholangitis (expected with biliary atresia)
Ascites (Hepatobiliary disorders) | 0 (0) | 1 (2) — Hospital admission for ascites management (expected with biliary atresia)
Bile leak (Hepatobiliary disorders) | 1 (1) | 0 (0) — Hospital admission for bile leak (can happen with biliary atresia)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pentoxifylline - Group 1 (Treatment Starts 3-5 Days After Kasai Portoenterostomy) (N=8) | Pentoxifylline - Group 2 (Patient Diagnosed Too Late for Kasai Portoenterostomy) (N=1)
ALT >2.5X baseline (Hepatobiliary disorders) | 1 (1) | 0 (0) — ALT levels 2.5X above level at Kasai portoenterostomy
Bc >2.5X baseline (Hepatobiliary disorders) | 0 (0) | 0 (0) — Conjugated bilirubin levels 2.5X above level at Kasai portoenterostomy
Platelets <150,000/ul (Blood and lymphatic system disorders) | 3 (3) | 1 (1) — Thrombocytopenia (sign of portal hypertension)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (5) — Vomiting from feeds and/or mediations, requiring change in feeding or medication regimen
Stopped medication before 12 week period (Product Issues) | 2 (2) | 0 (0) — Stopped medication before the study end period because of vomiting

LIMITATIONS AND CAVEATS:
Because of early termination, this study did not reach the target number of participants needed to achieve target power and statistically reliable results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-07): https://cdn.clinicaltrials.gov/large-docs/87/NCT01774487/Prot_SAP_000.pdf